CLINICAL TRIAL: NCT03909256
Title: NUTRI-HAB - A Randomised Controlled Trial on the Effect of a Targeted Residential Rehabilitation Program With a Focus on Eating Problems After Treatment for Head and Neck Cancer
Brief Title: NUTRI-HAB - Posttreatment Rehabilitation of Nutrition Impact Symptoms in Head and Neck Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: REHPA, The Danish Knowledge Centre for Rehabilitation and Palliative Care (Other); University of Southern Denmark (Other); University College Copenhagen (Other); Odense Patient Data Explorative Network (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Marianne Boll Kristensen, PhD student, Clinical dietitian, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 18/14847
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Head and Neck Cancer
Keywords: Rehabilitation; Nutrition impact symptoms; Quality of life
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The investigator will be blinded when performing the data analyses. Hence, data will be anonymised before analysis and the investigator will not know whether the group of subjects were allocated to the control or the intervention group.
  Results from blinded data analyses will be interpreted by project group before unblinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NUTRI-HAB (Experimental): The intervention group participates in a targeted rehabilitation program 'NUTRI-HAB' with a focus on eating problem after treatment for head and neck cancer. The program comprises:
  * a five day residential stay with patient education
  * a two day follow-up residential stay after 3 months
  * two telephone consultations with clinical dietitian between the two residential stays.
  Interventions: Other: NUTRI-HAB
- Control group (No Intervention): The control group receives no intervention other than usual care in the study period.
  After 3 months, the control group will be offered participation in the same residential rehabilitation program as the intervention group parcitipated in.

INTERVENTIONS:
Other: NUTRI-HAB — The rehabilitation program is a coordinated multidisciplinary effort involving several specialists e.g. clinical dietitians, nurses, physiotherapists, occupational therapists (responsible for dysphagia management in Denmark), psychologists and social workers.
  The program includes group sessions with patient education on how to handle the different aspects of living with eating problems and other late effects. Practical kitchen exercises, physical activity sessions and instruction in swallowing training are included. Individual counseling sessions with clinical dietitians and other health professionals (e.g. physicians) are offered depending on participants' needs.
  Participants stay at the premises and all meals throughout the day are served in the dining room or in the café. Foods of different textures and flavors are served to inspire participants and to allow them to experiment.
  Between the initial stay and follow-up participants are contacted twice by a clinical dietitian.
  Arms: NUTRI-HAB

SUMMARY:
The study is a randomised controlled trial that aims to test the effect of a residential rehabilitation program with a focus on eating problems after treatment in head and neck cancer survivors. The study will furthermore investigate whether selected nutrition screening and assessment tools can be used to identify head and neck cancer survivor who benefit from the program.

DETAILED DESCRIPTION:
This study is a randomised controlled trial with following objectives:

1. To test the effect of a targeted residential rehabilitation program with focus on the physical, psychological and social aspects of eating problems on body weight, health-related quality of life and physical function in curatively treated head and neck cancer survivors 1-5 years after completion of radiation therapy
2. To test whether a potential effect of the program is associated with/dependent of the participants' score in Scores Patient-Generated Subjective Global Assessment Short Form (PG-SGA-SF), Nutrition Risk Screening 2002 (NRS 2002) or M.D. Anderson Dysphagia Inventory (MDADI) at baseline

ELIGIBILITY:
Inclusion Criteria:

* Cancer of the larynx, pharynx or oral cavity
* Treatment with radiation therapy completed 1-5 years before inclusion
* Curatively treated
* Expression of interest in participating in the rehabilitation program in a preceding survey
* Self-reliant and no need for assistance with personal hygiene etc.

Exclusion Criteria:

* Active cancer disease at the time of recruitment
* Not being able to speak and understand Danish
* No permanent residence in Denmark

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Percentage change in body weight from baseline to follow up | Difference between measurements at baseline and at follow-up after 3 and 6 months
  Body weight will be measured with a calibrated scale at baseline and at follow up. Measurements will be performed by trained health professionals and standardised protocols will be followed. The change in percent will be calculated for each individual participant and be used as the primary outcome.

SECONDARY OUTCOMES:
Change in health-related quality of life (EORTC QLQ-C30) from baseline to follow up | Difference between measurements at baseline and at follow-up after 3 and 6 months
  Health-related quality of life (QOL) is measured using the generic EORTC QLQ-C30 questionnaire for cancer patients. Questionnaires will be scored according to EORTC's scoring manual, and changes from baseline to follow-up in the QOL-subscales will be calculated for each individual participant.
  The questionnaire consist of 30 items that are further divided into 15 subscales/items: a global health status/QOL scale; the functional scales: physical functioning, role functioning, emotional functioning, cognitive functioning, social functioning and the symptom scales/items: fatigue, nausea and vomiting, pain, dyspnoea, insomnia, appetite loss, constipation, diarrhoea, financial difficulties.
  All scales and single-item measures range in score from 0 to 100. A high score represents a higher response level. Thus a high score for a functional scale or global QOL represents a high level of functioning/QOL whereas a high score on a symptom scale represents a high level of symptoms.
Change in health-related quality of life (EORTC QLQ-H&N35) from baseline to follow up | Difference between measurements at baseline and at follow-up after 3 and 6 months
  Health-related quality of life (QOL) is measured using the questionnaire EORTC QLQ-H&N35 specific for head and neck cancer. Questionnaires will be scored according to EORTC's scoring manual, and changes from baseline to follow-up in the QOL-subscales will be calculated for each individual participant.
  The EORTC QLQ-H&N35 consists of 35 items that are further divided into the following symptom scales/items: pain, swallowing, sensory problems, speech problems, trouble with social eating, trouble with social contact, less sexuality, teeth, opening mouth, dry mouth, sticky saliva, coughing, felt ill, pain killers, nutritional supplements, feeding tube, weight loss, weight gain.
  All scales and single-item measures range in score from 0 to 100. A high score represents a higher response level. Thus a high score for symptom scale represents a high level of symptoms.
Change in health-related quality of life (EQ-5D-5L) from baseline to follow up | Difference between measurements at baseline and at follow-up after 3 and 6 months
  Health-related quality of life (QOL) is measured using EQ-5D-5L. Questionnaires will be scored according to manual, and changes from baseline to follow-up in the QOL-subscales will be calculated for each individual participant.
Percentage change in hand grip strength from baseline to follow up | Difference between measurements at baseline and at follow-up after 3 and 6 months
  Hand grip strength will be measured with a calibrated hand dynamometer at baseline and at follow up. Measurements will be performed by trained health professionals and standardised protocols will be followed. Three measurements will be performed for each participant and the mean will be calculated. The change in percent will be calculated for each individual participant.
Percentage change in '30 seconds sit-to-stand-test' from baseline to follow up | Difference between measurements at baseline and at follow-up after 3 and 6 months
  '30 seconds sit-to-stand-test' will be performed at baseline and follow-up. Measurements will be performed by trained health professionals and standardised protocols will be followed. The change in percent will be calculated for each individual participant.
Percentage change in '6 minutes walk test' from baseline to follow up | Difference between measurements at baseline and at follow-up after 3 and 6 months
  '6 minutes walk test' will be performed at baseline and follow-up. Measurements will be performed by trained health professionals and standardised protocols will be followed. The change in percent will be calculated for each individual participant.
Percentage change in mouth opening from baseline to follow up | Difference between measurements at baseline and at follow-up after 3 and 6 months
  Mouth opening will be measured at baseline and follow-up with TheraBite® Range-Of-Motion ROM Scale. The Therabite® ROM Scale is a disposable paper scale that measures the distance (in millimeters) between the upper and lower front teeth on maximal mouth opening. Lower values indicates trismus and increase indicates improvement. Measurements will be performed by trained health professionals and standardised protocols will be followed. The change in percent will be calculated for each individual participant.
Change in symptoms of anxiety and depression from baseline to follow up | Difference between measurements at baseline and at follow-up after 3 and 6 months
  Symptoms of anxiety and depression is measured with the Hospital Anxiety and Depression Scale

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Dorthe Zwisler, Professor, Study Director — REHPA, The Danish Knowledge Centre for Rehabilitation and Palliative Care
Locations (1):
- REHPA, The Danish Knowledge Centre for Rehabilitation and Palliative Care, Nyborg, Denmark

IPD SHARING:
Plan to Share IPD: No
Within the confines of Danish legislation, anonymised data from the trial will be available for other researchers upon reasonable request when results have been published.

REFERENCES:
- [Derived] Kristensen MB, Wessel I, Beck AM, Dieperink KB, Mikkelsen TB, Moller JK, Zwisler AD. Rationale and design of a randomised controlled trial investigating the effect of multidisciplinary nutritional rehabilitation for patients treated for head and neck cancer (the NUTRI-HAB trial). Nutr J. 2020 Mar 17;19(1):21. doi: 10.1186/s12937-020-00539-7. PMID 32183835